CLINICAL TRIAL: NCT00939185
Title: Compliance And Safety Study In Children With Upper And Lower Respiratory Tract Infections
Acronym: COMPAS
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: A0661182
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Results first posted 2010-03-18 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Respiratory Tract Infections
Keywords: Compliance and Safety Study in Children with Upper and Lower Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections; Patient Compliance | interventions — Azithromycin

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Azithromycin group
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — Zithromax was dispensed according to the Summary of Product Characteristics (SPC) as either a tablet or suspension. Zithromax was administered as a total dose of 30 mg/kg which was given as single daily doses of 10 mg/kg for 3 days, or as a 5 day dose starting with 10 mg/kg on Day 1, then 5 mg/kg on Days 2-5.
  Other Names: Zithromax

SUMMARY:
The objective of this study was to obtain data on the safety, tolerability and compliance with Zithromax in children with bacterial infections of the upper and lower respiratory tract.

DETAILED DESCRIPTION:
Patients were recruited from the outpatient departments of the participating sites/hospitals/clinics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with respiratory tract infections that received azithromycin according to the approved SPC as this was a non-interventional study.

Exclusion Criteria:

* According to the approved Summary of Product Characteristics (SPC) for Azithromycin as this was a non interventional study.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: ZITHROMAX® administration will be considered in children / adolescents from the first year of life up to 14 years old with the following diagnoses: Acute otitis media, Sinusitis, Pharyngitis/tonsillitis, Pneumonia, Bronchitis.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2007-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661182&StudyName=Compliance%20And%20Safety%20Study%20In%20Children%20With%20Upper%20And%20Lower%20Respiratory%20Tract%20Infections

RESULTS

PARTICIPANT FLOW:
Groups:
- Azithromycin: The total dose of 30 mg/kg could have been given as a single daily dose of 10 mg/kg daily for 3 days, or given over 5 days with a single daily dose of 10 mg/kg on Day 1, then 5 mg/kg on Days 2-5. For pediatric streptococcal pharyngitis, azithromycin could have been given as a single dose of 10 mg/kg or 20 mg/kg for 3 days; with a maximum daily dose of 500 mg. For children with acute otitis media, a single dose of 30 mg/kg could have been given.
Period: Overall Study
Arm/Group | Azithromycin
Started | 400
Received Treatment | 390
Completed | 375
Not Completed | 25
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 6
Not completed — Other | 3
Not completed — Withdrawal by Subject | 2
Not completed — Randomized But Did Not Receive Treatment | 10

BASELINE CHARACTERISTICS:
Arm/Group | Azithromycin
Number analyzed (Participants) | 390
Age, Customized [Number; unit: participants]
  Birth to 1 month | 2
  > 1 month to 2 years | 82
  > 2 years to 12 years | 292
  > 12 years to 18 years | 10
  > 18 years | 0
  Unspecified | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167
  Male | 223

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events (AEs)
Description: All observed or volunteered AEs regardless of suspected causal relationship to the investigational product(s) were reported.
Time Frame: 3 to 7 days after receiving treatment
Population: Safety population = Those subjects who were known to have received at least one dose of the study treatment. Subjects who were dispensed study treatment and immediately lost to follow-up were not included among those known to have been dosed.
Measure: Number; unit: participants
Arm/Group | Azithromycin
Number analyzed (Participants) | 390
participants | 27

2. Secondary Outcome: Number of Subjects Who Withdrew From the Study
Time Frame: 3 to 7 days after receiving treatment
Population: Safety Population. Please refer to the participant flow and AE sections for results pertaining to tolerability.
Measure: Number; unit: participants
Arm/Group | Azithromycin
Number analyzed (Participants) | 0

3. Secondary Outcome: Compliance
Description: Compliance was assessed by the following questions: Question 1: "Were the pediatrician's instructions during the treatment phase followed (i.e. dose, frequency and number of days)?"; Question 2: "Was it easy to understand your pediatrician's instructions regarding treatment?"; and Question 3: "Was the administration of this drug easier than any other previously used drug?" Patients could answer either "yes", "no", or "Not applicable (NA)".
Time Frame: 3 to 7 days after receiving treatment
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Azithromycin
Number analyzed (Participants) | 390
participants
  Question 1: Yes | 370
  Question 1: No | 13
  Question 1: NA | 6
  Question 1: Missing | 1
  Question 2: Yes | 374
  Question 2: No | 9
  Question 2: NA | 6
  Question 2: Missing | 1
  Question 3: Yes | 356
  Question 3: No | 22
  Question 3: NA | 11
  Question 3: Missing | 1

4. Secondary Outcome: Time Reported for a Patient Being Consulted and Diagnosed From the Moment He/She Entered the Hospital
Description: Time of exam completion minus the start time of the examination.
Time Frame: Day 1
Population: Safety population
Measure: Median (Full Range); unit: minutes
Arm/Group | Azithromycin
Number analyzed (Participants) | 398
minutes | 20 [5 to 585]

ADVERSE EVENTS:
Arm/Group | Azithromycin
Serious Adverse Events (participants affected / at risk) | 0/390
Other Adverse Events (participants affected / at risk) | 27/390
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azithromycin (N=390)
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Chest pain (General disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Anxiety (Psychiatric disorders) | 2
Diaphragmalgia (Respiratory, thoracic and mediastinal disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Only 1 subject received tablet; therefore, no suspension versus tablet efficacy data is displayed as initially planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.